CLINICAL TRIAL: NCT02606136
Title: Trial of Pamrevlumab (FG-3019), a Monoclonal Antibody to Connective Tissue Growth Factor, in Non-Ambulatory Subjects With Duchenne Muscular Dystrophy
Brief Title: Trial of Pamrevlumab (FG-3019), in Non-Ambulatory Participants With Duchenne Muscular Dystrophy (DMD)
Acronym: MISSION
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-3019-079; 2023-000321-80 (EudraCT Number)
Record Dates: First submitted 2015-11-04; First posted 2015-11-17 (Estimated); Results first posted 2021-12-30 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne; muscular; dystrophy; DMD; non-ambulatory
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — pamrevlumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Pamrevlumab (Experimental): Participants will receive pamrevlumab 35 milligrams (mg)/kilogram (kg) by intravenous (IV) infusion every 2 weeks for a minimum of 104 weeks. Participants who complete the main study, will continue to receive pamrevlumab 35 mg/kg by IV infusion every 2 weeks for a minimum of up to 208 weeks in the OLE.
  Interventions: Drug: Pamrevlumab

INTERVENTIONS:
Drug: Pamrevlumab — Pamrevlumab, 10 milligrams (mg)/milliliter (mL), single dose vials
  Other Names: Monoclonal Antibody to Connective tissue growth factor (CTGF), FG-3019

SUMMARY:
This is a Phase 2, open-label, single arm trial of pamrevlumab (FG-3019) to estimate pamrevlumab's safety and efficacy in non-ambulatory participants with DMD.

DETAILED DESCRIPTION:
The study will include a screening period, main study period, open-label extension (OLE) period, and follow-up period 4 weeks after the last dose. All participants who complete the main portion of the study for a minimum of 104 weeks (2 years) will be rolled over to an OLE for up to an additional 208 weeks (4 years).

ELIGIBILITY:
Inclusion Criteria:

* Written consent/assent by participant and/or legal guardian as per regional and/or institutional review board (IRB) requirements
* Non-ambulatory
* Brooke Score for Arms and Shoulders ≤5
* Diagnosis of DMD by medical history and confirmed Duchenne mutation in available genetic testing using a validated genetic test
* Able to perform spirometry
* Able to undergo cardiac and extremity (upper arm) MRI
* Percent predicted FVC between 40 and 90, inclusive
* At least one historical ppFVC predicted value within 18 months of baseline
* Left ventricular ejection fraction ≥ 45% as determined by cardiac MRI at screening or within 3 months prior to Day 0
* Participants currently receiving heart failure cardiac medications (for example, angiotensin converting enzyme inhibitors, angiotensin-receptor blockers, and beta-blockers) must achieve a stable regimen for at least 3 months prior to screening
* On a stable dose of corticosteroids for a minimum of 6 months prior to screening with no substantial change in dosage for a minimum of 3 months (except for adjustments for changes in body weight) prior to screening and no foreseen change in corticosteroid use during the course of study participation
* Received pneumococcal vaccine and is receiving annual influenza vaccinations
* Adequate renal function: cystatin C ≤1.4 mg/liter (L)
* Adequate hematological function

  1. Platelets >100,000/microliter (μL)
  2. Hemoglobin >12 grams (g)/deciliter (dL)
  3. Absolute neutrophil count >1500/μL
* Adequate hepatic function

  1. No history or evidence of liver disease
  2. Gamma glutamyl transferase (GGT) ≤3 x upper limit of normal (ULN)
  3. Total bilirubin ≤1.5 x ULN
* If sexually active, will use medically accepted contraceptives during participation in the study and for 3 months after the last dose of study drug

Exclusion Criteria:

* Requires ≥16 hours continuous ventilation
* Prior or ongoing medical condition that, in the investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of 156 weeks of treatment and follow-up would be completed, or could impair the assessment of study results
* Anticipated spine surgery within 156 weeks
* Severe uncontrolled heart disease, including any of the following:

  1. Need for intravenous diuretics or inotropic support within 3 months prior to screening
  2. Hospitalization for a heart failure exacerbation or arrhythmia in last 3 months
* Arrhythmia requiring anti-arrhythmic therapy
* Hospitalization due to respiratory failure in the last 6 weeks
* Poorly controlled asthma or underlying lung disease such as bronchopulmonary dysplasia
* Known or suspected active hepatitis B or C or history of human immunodeficiency virus (HIV)
* Body mass index (BMI) ≥40 kilograms (kg)/square meter (m^2) or weight >117 kg
* Exposure to another investigational drug or another approved product for DMD (for example, eteplirsen or golodirsen) within 28 days prior to start of study treatment
* Exposure to another investigational drug or another approved product for DMD (e.g. eteplirsen) within 28 days prior to start of study treatment (or 5 half-lives of the product whichever is longer) prior to first screening visit with the exception of deflazacort. Use of deflazacort, if regarded by the principal investigator as standard of care, is allowed.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2023-08-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California San Francisco - Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rare Disease Research, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Shriner's Hospital for Children - Portland, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center Ambulatory Care Pavilion, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rayego-Mateos S, Morgado-Pascual JL, Lavoz C, Rodrigues-Diez RR, Marquez-Exposito L, Tejera-Munoz A, Tejedor-Santamaria L, Rubio-Soto I, Marchant V, Ruiz-Ortega M. CCN2 Binds to Tubular Epithelial Cells in the Kidney. Biomolecules. 2022 Feb 3;12(2):252. doi: 10.3390/biom12020252. PMID 35204752

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who completed the main portion of the study for a minimum of 104 weeks (2 years) were rolled over to an open-label extension (OLE) for up to an additional 208 weeks (4 years). Some participants remained in the main study for up to 206 weeks before rolling over to the OLE.
Groups:
- Pamrevlumab: Participants received pamrevlumab 35 milligrams (mg)/kilogram (kg) by intravenous (IV) infusion every 2 weeks for a minimum of 104 weeks in the main study. Participants who completed the main study, continued to receive pamrevlumab 35 mg/kg by IV infusion every 2 weeks for a minimum of up to 208 weeks in the OLE.
Period: Main Study (104 Weeks)
Arm/Group | Pamrevlumab
Started | 21
Received at Least 1 Dose of Study Drug | 21
Completed | 15
Not Completed | 6
Not completed — Participant/Legal Guardian Decision | 5
Not completed — Withdrawal by Subject | 1
Period: OLE (Up to 208 Weeks)
Arm/Group | Pamrevlumab
Started | 15
Received at Least 1 Dose of Study Drug | 15
Completed | 0
Not Completed | 15
Not completed — Participant/Legal Guardian Decision | 1
Not completed — Sponsor Decision to Terminate Study | 14

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who enrolled in the study.
Groups:
- Pamrevlumab: Participants received pamrevlumab 35 mg/kg by IV infusion every 2 weeks for a minimum of 104 weeks in the main study. Participants who completed the main study, continued to receive pamrevlumab 35 mg/kg by IV infusion every 2 weeks for a minimum of up to 208 weeks in the OLE.
Arm/Group | Pamrevlumab
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.99 (3.277)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Percent Predicted Forced Vital Capacity (ppFVC) [Mean (Full Range); unit: percentage of predicted FVC] — FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC was the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted FVC is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FVC = (observed value)/(predicted value) * 100%.
  percentage of predicted FVC | 54.15 [29.1 to 70.7]
Percent Predicted Peak Expiratory Flow (PEF) [Mean (Full Range); unit: percentage of predicted PEF] — Percent predicted PEF is a measure of the maximal or peak flow produced during an exhalation with maximal effort and, as such, is the most effort-dependent measure of lung function.
  percentage of predicted PEF | 54.66 [37.9 to 82.7]
Percent Predicted Forced Expiratory Volume at 1 Second (ppFEV1) [Mean (Full Range); unit: percentage of predicted FEV1] — FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Predicted FEV1 is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FEV1= (observed value)/(predicted value) * 100%.
  percentage of predicted FEV1 | 53.815 [29.24 to 73.35]
Left Ventricular Ejection Fraction Percentage (LVEF%) [Mean (Full Range); unit: percentage of LVEF] — LVEF% is an important measure of cardiac function. LVEF is a fraction of blood (in percent) pumped out of the left ventricle of the heart (the main pumping chamber).
  percentage of LVEF | 56.992 [41.03 to 73.81]
Performance of Upper Limb (PUL) Total Score [Mean (Full Range); unit: unit on a scale] — The PUL module is an observer-administered performance battery of upper extremity mobility tasks for the shoulder (upper, 6 items: maximum score = 12), elbow (middle, 9 items: maximum score = 17) and wrist/hand (distal, 7 items: maximum score = 13). Higher scores of each item indicate higher level of function. Total score was calculated by adding the 3 level scores, with a maximum global score of 42 (total score range = 0-42; with higher score indicating better outcome).
  unit on a scale | 24.4 [13 to 41]
Pinch Strength, as Measured by Hand Held Myometry (HHM) [Mean (Full Range); unit: newton] — The HHM was used to measure distal upper arm strength (pinch strength). Data has been presented by dominant and non-dominant hand.
  newton
    Dominant Pinch Best Result | 17.003 [0 to 45.1]
    Non-Dominant Pinch Best Result | 16.607 [0 to 47.1]
Grip Strength by Hand, as Measured by HHM [Mean (Full Range); unit: newton] — The HHM was used to measure distal upper arm strength (grip strength). Data has been presented by dominant and non-dominant hand.
  newton
    Dominant Grip Best Result | 45.861 [3 to 142.2]
    Non-Dominant Grip Best Result | 41.977 [2 to 104.9]
Cardiac Fibrosis Score (Scar Mass), as Measured by Magnetic Resonance Imaging (MRI) [Mean (Full Range); unit: grams] — Population: 'Number analyzed' signifies participants evaluable for this parameter.
  grams
    number analyzed (Participants) | 20
    (all) | 24.100 [0.44 to 76.09]
Upper Arm (Biceps Brachii MRI) Muscle Fat and Fibrosis Score [Mean (Full Range); unit: unit on a scale] — T2-mapping with MRI was conducted to measure upper arm muscle fibrosis and fat in the biceps brachii muscle. Population: 'Number analyzed' signifies participants evaluable for this parameter.
  unit on a scale
    number analyzed (Participants) | 12
    (all) | 8.01 [3.9 to 17.2]
Fat Fraction Percentage (%F), as Measured by MRI [Mean (Full Range); unit: percentage of fat] — Population: 'Number analyzed' signifies participants evaluable for this parameter.
  percentage of fat
    number analyzed (Participants) | 9
    (all) | 22.07 [4 to 32.6]

OUTCOME MEASURES:

1. Primary Outcome: Annual Change From Baseline in Percent Predicted Forced Vital Capacity (ppFVC) at Week 104
Description: FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC was the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted FVC is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FVC = (observed value)/(predicted value) * 100%. Analysis was done using a random coefficient model (RCM), which included visit in years (as a continuous variable), and baseline efficacy as fixed effects, the intercept and the linear slope of visit as random effect, and individual participants as participant effect.
Time Frame: Baseline, Week 104
Population: ITT population included all participants who enrolled in the study.
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted FVC
Groups:
- Pamrevlumab: Participants received pamrevlumab 35 mg/kg by IV infusion every 2 weeks for a minimum of 104 weeks.
Arm/Group | Pamrevlumab
Number analyzed (Participants) | 21
percentage of predicted FVC | -4.17 (0.655)

2. Secondary Outcome: Change From Baseline in Percent Predicted Forced Expiratory Volume at 1 Second (ppFEV1) at Week 104
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Predicted FEV1 is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FEV1= (observed value)/(predicted value) * 100%. Analysis was done using an RCM, which included visit in years (as a continuous variable), and baseline efficacy as fixed effects, the intercept and the linear slope of visit as random effect, and individual participants as participant effect.
Time Frame: Baseline, Week 104
Population: ITT population included all participants who enrolled in the study.
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted FEV1
Arm/Group | Pamrevlumab
Number analyzed (Participants) | 21
percentage of predicted FEV1 | -8.32 (1.217)

3. Secondary Outcome: Change From Baseline in Percent Predicted Peak Expiratory Flow (PEF) at Week 104
Description: Percent predicted PEF is a measure of the maximal or peak flow produced during an exhalation with maximal effort and, as such, is the most effort-dependent measure of lung function. Analysis was done using an RCM, which included visit in years (as a continuous variable), and baseline efficacy as fixed effects, the intercept and the linear slope of visit as random effect, and individual participants as participant effect.
Time Frame: Baseline, Week 104
Population: ITT population included all participants who enrolled in the study.
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted PEF
Arm/Group | Pamrevlumab
Number analyzed (Participants) | 21
percentage of predicted PEF | -7.13 (2.313)

4. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction Percentage (LVEF%) at Week 104
Description: LVEF% is an important measure of cardiac function. LVEF is a fraction of blood (in percent) pumped out of the left ventricle of the heart (the main pumping chamber). Analysis was done using an RCM, which included visit in years (as a continuous variable), and baseline efficacy as fixed effects, the intercept and the linear slope of visit as random effect, and individual participants as participant effect.
Time Frame: Baseline, Week 104
Population: ITT population included all participants who enrolled in the study.
Measure: Least Squares Mean (Standard Error); unit: percentage of LVEF
Arm/Group | Pamrevlumab
Number analyzed (Participants) | 21
percentage of LVEF | -2.73 (1.651)

5. Secondary Outcome: Change From Baseline in Performance of Upper Limb (PUL) Total Score at Week 104
Description: The PUL module is an observer-administered performance battery of upper extremity mobility tasks for the shoulder (upper, 6 items: maximum score = 12), elbow (middle, 9 items: maximum score = 17) and wrist/hand (distal, 7 items: maximum score = 13). Higher scores of each item indicate higher level of function. Total score was calculated by adding the 3 level scores, with a maximum global score of 42 (total score range = 0-42; with higher score indicating better outcome). Analysis was done using an RCM, which included visit in years (as a continuous variable), and baseline efficacy as fixed effects, the intercept and the linear slope of visit as random effect, and individual participants as participant effect.
Time Frame: Baseline, Week 104
Population: ITT population included all participants who enrolled in the study.
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Pamrevlumab
Number analyzed (Participants) | 21
unit on a scale | -4.14 (0.651)

6. Secondary Outcome: Change From Baseline in Grip Strength by Hand, as Measured by Hand Held Myometry (HHM) at Week 104
Description: The HHM was used to measure distal upper arm strength (grip strength). Data has been presented by dominant and non-dominant hand. Analysis was done using an RCM, which included visit in years (as a continuous variable), and baseline efficacy as fixed effects, the intercept and the linear slope of visit as random effect, and individual participants as participant effect.
Time Frame: Baseline, Week 104
Population: ITT population included all participants who enrolled in the study.
Measure: Least Squares Mean (Standard Error); unit: newton
Arm/Group | Pamrevlumab
Number analyzed (Participants) | 21
newton
  Dominant Grip Best Result | -2.52 (3.610)
  Non-Dominant Grip Best Result | -1.31 (3.591)

7. Secondary Outcome: Change From Baseline in Pinch Strength, as Measured by HHM at Week 104
Description: The HHM was used to measure distal upper arm strength (pinch strength). Data has been presented by dominant and non-dominant hand. Analysis was done using an RCM, which included visit in years (as a continuous variable), and baseline efficacy as fixed effects, the intercept and the linear slope of visit as random effect, and individual participants as participant effect.
Time Frame: Baseline, Week 104
Population: ITT population included all participants who enrolled in the study.
Measure: Least Squares Mean (Standard Error); unit: newton
Arm/Group | Pamrevlumab
Number analyzed (Participants) | 21
newton
  Dominant Pinch Best Result | -4.24 (1.547)
  Non-Dominant Pinch Best Result | -3.46 (1.378)

8. Secondary Outcome: Change From Baseline in Cardiac Fibrosis (Scar Mass), as Measured by Magnetic Resonance Imaging (MRI) at Week 104
Description: Cardiac MRI was used to assess the cardiac fibrosis by detecting the presence of late gadolinium enhancement (LGE), a marker for myocardial fibrosis. Analysis was done using an RCM, which included visit in years (as a continuous variable), and baseline efficacy as fixed effects, the intercept and the linear slope of visit as random effect, and individual participants as participant effect.
Time Frame: Baseline, Week 104
Population: ITT population included all participants who enrolled in the study. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Pamrevlumab
Number analyzed (Participants) | 20
grams | 3.74 (4.475)

9. Secondary Outcome: Change From Baseline in Upper Arm (Biceps Brachii MRI) Muscle Fat and Fibrosis Score, as Measured by MRI at Week 104
Description: T2-mapping with MRI was conducted to measure upper arm muscle fibrosis and fat in the biceps brachii muscle. Analysis was done using an RCM, which included visit in years (as a continuous variable), and baseline efficacy as fixed effects, the intercept and the linear slope of visit as random effect, and individual participants as participant effect. The visual score for muscle fat and fibrosis will be assessed using a modified 5-point Mercuri score in which 0 = normal muscle appearance and 5 = complete replacement of muscle by connective tissue and fat, where a lower score indicated visually healthier muscle. Change from baseline was calculated as the score at Week 104 - the score at baseline.
Time Frame: Baseline, Week 104
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: unit on scale
Arm/Group | Pamrevlumab
Number analyzed (Participants) | 12
unit on scale | -2.22 (1.088)

10. Secondary Outcome: Change From Baseline in Fat Fraction Percentage (%F), as Measured by MRI at Week 104
Description: Analysis was done using an RCM, which included visit in years (as a continuous variable), and baseline efficacy as fixed effects, the intercept and the linear slope of visit as random effect, and individual participants as participant effect.
Time Frame: Baseline, Week 104
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: percentage of fat
Arm/Group | Pamrevlumab
Number analyzed (Participants) | 9
percentage of fat | 4.49 (2.030)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 210
Description: Safety population included participants who received at least one dose of study drug.
Groups:
- Main Study: Pamrevlumab: Participants received pamrevlumab 35 mg/kg by IV infusion every 2 weeks for a minimum of 104 weeks.
- OLE: Pamrevlumab: Participants who completed the main study, continued to receive pamrevlumab 35 mg/kg by IV infusion every 2 weeks for a minimum of up to 208 weeks in the OLE.
Arm/Group | Main Study: Pamrevlumab | OLE: Pamrevlumab
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/15
Serious Adverse Events (participants affected / at risk) | 6/21 | 5/15
Other Adverse Events (participants affected / at risk) | 21/21 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Pamrevlumab (N=21) | OLE: Pamrevlumab (N=15)
Food poisoning (Gastrointestinal disorders) | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Retinal exudates (Eye disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Catheter site abscess (Infections and infestations) | 0 | 1
Pilonidal disease (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Pamrevlumab (N=21) | OLE: Pamrevlumab (N=15)
Palpitations (Cardiac disorders) | 3 | 0
Ear pain (Ear and labyrinth disorders) | 3 | 2
Cataract (Eye disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 10 | 2
Nausea (Gastrointestinal disorders) | 7 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Pyrexia (General disorders) | 8 | 1
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 3
Vaccination site pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 1 | 3
Medical device site rash (General disorders) | 0 | 2
Hypersensitivity (Immune system disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 11 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 3
Sinusitis (Infections and infestations) | 3 | 0
Influenza (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 2 | 2
Bone contusion (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 2
Sunburn (Injury, poisoning and procedural complications) | 1 | 1
Cystatin C increased (Investigations) | 2 | 1
Weight decreased (Investigations) | 2 | 0
Bone density decreased (Investigations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Headache (Nervous system disorders) | 14 | 4
Dizziness (Nervous system disorders) | 3 | 0
Migraine (Nervous system disorders) | 2 | 1
Sinus headache (Nervous system disorders) | 2 | 0
Fine motor skill dysfunction (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 1
Depression (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Cardiac dysfunction (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Chalazion (Eye disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 4
Ear infection (Infections and infestations) | 0 | 2
Fungal infection (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 2
Infected cyst (Infections and infestations) | 0 | 1
Pilonidal disease (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Skin candida (Infections and infestations) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuromuscular scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen. The investigator can only publish after the multisite consortium publishes (or tries to publish and fails). FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT02606136/Prot_002.pdf
  • Statistical Analysis Plan (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT02606136/SAP_003.pdf